CLINICAL TRIAL: NCT02934867
Title: Out of Hospital Cardiac Arrest: Cluster Randomized Trial Assessing the Survival Impact of Phone Advice Delivered by Medical Call Center
Brief Title: Out of Hospital Cardiac Arrest: Trial Assessing the Survival Impact of Phone Advice
Acronym: CONTAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Central Hospital, Nancy, France (Other); University Hospital, Metz (Unknown); University Hospital, Strasbourg, France (Other); Reims University hospital (Other); Centre Hospitalier de Lons Le Saunier (Unknown); Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other); Centre Hospitalier de Colmar (Other); Centre Hospitalier de Troyes (Other); Centre Hospitalier de Chalon sur Saône (Unknown); Centre Hospitalier Universitaire de Nīmes (Other); Nantes University Hospital (Other); University Hospital, Bordeaux (Other); Hospices Civils de Lyon (Other); Poitiers University Hospital (Other); University Hospital, Angers (Other Government); University Hospital, Orléans (Unknown); Centre Hospitalier de Montauban (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONTAC R/2015/50
Record Dates: First submitted 2016-07-26; First posted 2016-10-17 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2020-01

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTARM (Experimental): Protocol phone advice
  Interventions: Other: Protocol phone advice
- CONTHAB (Other): Usual phone advice
  Interventions: Other: Usual phone advice

INTERVENTIONS:
Other: Protocol phone advice — Protocol phone advice
  Arms: CONTARM
Other: Usual phone advice — Usual phone advice
  Arms: CONTHAB

SUMMARY:
Medical call center have no phone advice protocol within out of hospital cardiac arrest in France. The purpose of the present study is to compare a group of patients with protocol phone advice delivered by the dispatchers ("CONTARM" group) versus usual phone advice ( "CONTHAB" group). Comparison will be performed on survival to seven days. The hypothesis is that CONTARM group has an higher survival at seven days. A second goal is to measure the survival to 15 and 30 days. The trial is randomized, controlled and will include 2600 patients. The patients will be enrolled in 19 hospitals in France.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* initial call to 15
* out of hospital cardiac arrest
* patient proximity to witness

Exclusion Criteria:

* first aid professionals on site
* rigor mortis
* location not allowing resuscitation
* inability to realize actions or misunderstanding
* no flow > 5 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
7 days survival | 7 days
  7 days survival

SECONDARY OUTCOMES:
15 and 30 days survival | 15 and 30 days
  15 and 30 days survival
Assessment of compliance of phone advice | 7 days
  Listening of phone bands to measure compliance of phone advice protocol :
  * good frequency of chest compression. Binary variable (Yes or Not)
  * good depth of chest compression. Binary variable (Yes or Not)
  * good patient positioning. Binary variable (Yes or No).
30 days neurological status | 30 days
  Cerebral performance categories scale is counting with medical file

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CH Châlon sur Saône, Châlon Sur Saône
  - CH Colmar, Colmar
  - CHU Dijon, Dijon
  - CH Lons Le Saunier, Lons-le-Saunier
  - CHU Lyon, Lyon
  - CHU Metz, Metz
  - CH Montauban, Montauban
  - CH Mulhouse, Mulhouse
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nîmes, Nîmes
  - CH Orléans, Orléans
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Strasbourg, Strasbourg
  - CH Troyes, Troyes

REFERENCES:
- [Background] Berg RA, Hemphill R, Abella BS, Aufderheide TP, Cave DM, Hazinski MF, Lerner EB, Rea TD, Sayre MR, Swor RA. Part 5: adult basic life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S685-705. doi: 10.1161/CIRCULATIONAHA.110.970939. PMID 20956221
- [Background] Nolan JP, Soar J, Zideman DA, Biarent D, Bossaert LL, Deakin C, Koster RW, Wyllie J, Bottiger B; ERC Guidelines Writing Group. European Resuscitation Council Guidelines for Resuscitation 2010 Section 1. Executive summary. Resuscitation. 2010 Oct;81(10):1219-76. doi: 10.1016/j.resuscitation.2010.08.021. No abstract available. PMID 20956052
- [Background] Koster RW, Baubin MA, Bossaert LL, Caballero A, Cassan P, Castren M, Granja C, Handley AJ, Monsieurs KG, Perkins GD, Raffay V, Sandroni C. European Resuscitation Council Guidelines for Resuscitation 2010 Section 2. Adult basic life support and use of automated external defibrillators. Resuscitation. 2010 Oct;81(10):1277-92. doi: 10.1016/j.resuscitation.2010.08.009. No abstract available. PMID 20956051
- [Background] Desmettre T, Jenvrin J, Freysz M, Nace L, Puyraveau M, Berthier F, Dreyfus P, Philippe MH, Labourey JM, Capellier G. Drug prescription at the medical call center. Ann. Fr. Med. Urgence (2013) 3:14-19.
- [Background] Sigaux A, Jonquet S, Puyraveau M, Bretillot L, Labourey JM, Capellier G, Desmettre T. Evaluation of phone advice delivered by a medical call center in case of cardiac arrest. Ann. Fr. Med. Urgence (2014) 4:11-17.